CLINICAL TRIAL: NCT00656955
Title: Follow-up of Kidney Cancer Patients From the Central European Multicenter Case-Control Study
Brief Title: Follow-Up Study of Kidney Cancer Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908107; 08-C-N107
Record Dates: First submitted 2008-04-11; First posted 2008-04-14 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Renal Cancer
Keywords: Kidney Cancer; Molecular Epidemiology; Survival; Occupational Exposures; Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal cancer patients: Renal cancer patients

SUMMARY:
Background:

In Central Europe, mortality rates for kidney cancers are higher and survival rates are lower than in the United States and Western Europe overall.

The Central and Eastern European Renal Cancer Case-Control Study (CEERCC), completed in 2002, offers an opportunity to identify determinants that predict 5-year survival among kidney cancer patients.

Objectives:

To assess disease recurrence and progression among former participants in the CEERCC.

To investigate the effect of genetics, lifestyle factors, medical conditions, occupation and diet on the outcome of kidney cancer patients in Europe.

Eligibility:

Former participants or next-of-kin of former participants in the CEERCC study.

Design:

Participants or their next-of-kin are interviewed for 60 minutes and are requested permission to collect relevant information from their or their family member s hospital and cancer registry records.

DETAILED DESCRIPTION:
Previously we proposed to conduct a follow-up study of kidney cancer in the high risk region of Central and Eastern Europe. This study was conducted through the follow-up of a group of patients with kidney cancer, that were previously enrolled in the study entitled, Occupation, Genetic Susceptibility Kidney Cancer: Central European Case-Controls Study, PI Dr. Wong-Ho Chow, OEEB, DCEG, NCI, protocol No 01-C-NO63, a study for which field work and data analyses of the case control study were completed. We had originally planned to conduct the follow-up study in seven centers in four countries, including Romania, Poland, Russia, and the Czech Republic. In each center, cancer-related information was to be extracted from vital statistics, cancer registry, and/or medical records. For deceased patients, next-of-kin were to be interviewed using a brief questionnaire.

A pilot study was conducted to determine the feasibility of collecting survival information including 5-year survival status, date of death, cause of death, and date of last follow-up if alive from 220 cases across the seven collaborating centers. The feasibility of extracting additional data including surgical and medical treatment procedures used to treat primary disease, the recurrence and progression of primary disease was also determined. However, based on results obtained from the pilot study, we determined that it is feasible to collect follow-up data from kidney cancer cases from four centers in the Czech Republic and one center in both Poland and Russia.

Medical records/archives for Romanian cases were located in hospitals that were completely destroyed during reconstruction therefore, it was impossible to collect any information from this subset of patients. Exclusion of these records will not affect study power since most of the cases were from the Czech Republic. The objective of our proposed study remains the same:( 1) to assess the 5-year survival status of kidney cancer patients in the Central and Easter European Renal Cell Carcinoma Study; (2) to examine prevalence of recurrent disease and progression; (3) to investigate additional patient-tumor-and genetic determinant of 5-year survival in cases.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this study, patients needed to have participated as a histologically confirmed renal cancer case in the previous case-control study entitled Central European Renal Cancer Case-Control (CEERCC) Study which was completed in 2002.

EXCLUSION CRITERIA:

Children less than 18 are not eligible to participate in this study because there were no kidney cancer cases observed in the CEERCC Study that were less than 18 years of age.

American Indian/Alaskan Native, Asian, Black or African American, Hispanic or Latino, and Native Hawaiian or Pacific Islander.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal cancer patients
Sampling Method: Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2008-04-17 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Survival | Months of cancer-free survival
  Cause-specific and overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Purdue, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- Czechia (2):
  - Dept of Cancer Epidemioology Genetics, Brno, CZ, Brno
  - Olomouc University, Olomouc
- National Institute of Occupational Medicine, Lodz, Poland, Lodz, Poland